CLINICAL TRIAL: NCT03956238
Title: Integrating Alcohol Myopia and Objectification to Understand Sexual Assault
Brief Title: Alcohol Myopia, Objectification, and Sexual Assault
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18599; R01AA025090 (NIH)
Record Dates: First submitted 2019-05-02; First posted 2019-05-20 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Alcoholic Intoxication
Keywords: Alcohol intoxication; Alcohol use; Drinking; Sexual assault; Sexual violence; Aggression; Attention; Victimization; Public health
MeSH Terms: conditions — Alcoholic Intoxication; Alcohol Drinking; Aggression | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Males and Alcohol Intoxication (Experimental): Men assigned to alcohol intoxication arm (target BAC .08%)
  Interventions: Behavioral: Alcohol intoxication
- Males and Placebo Control (Placebo Comparator): Men assigned to placebo control arm
  Interventions: Behavioral: Alcohol intoxication
- Females and Alcohol Intoxication and Objectifying Gazes (Experimental): Women assigned to alcohol intoxication arm (target BAC .08%) and objectifying gazes arm
  Interventions: Behavioral: Alcohol intoxication; Behavioral: Objectification
- Females and Alcohol Intoxication and Eye Gazes (Experimental): Women assigned to alcohol intoxication arm (target BAC .08%) and eye gazes arm
  Interventions: Behavioral: Alcohol intoxication; Behavioral: Objectification
- Females and Placebo Control and Objectifying Gazes (Experimental): Women assigned to placebo control arm and objectifying gazes arm
  Interventions: Behavioral: Alcohol intoxication; Behavioral: Objectification
- Females and Placebo Control and Eye Gazes (Placebo Comparator): Women assigned to placebo control arm and eye gazes arm
  Interventions: Behavioral: Alcohol intoxication; Behavioral: Objectification

INTERVENTIONS:
Behavioral: Alcohol intoxication — Men and women assigned to moderate alcohol dose condition (target BAC .08%) or placebo control condition with NIAAA approved alcohol administration procedures
Behavioral: Objectification — Women assigned to objectifying gazes condition or eye contact control condition
  Arms: Females and Alcohol Intoxication and Eye Gazes; Females and Alcohol Intoxication and Objectifying Gazes; Females and Placebo Control and Eye Gazes; Females and Placebo Control and Objectifying Gazes

SUMMARY:
The present project integrates previous research on factors associated with alcohol-involved sexual assault, with research on how intoxication alters attention and social perceptions in ways that increase the risk of sexual aggression and victimization. Specifically, this project examines whether alcohol intoxication on the part of a male perpetrator impairs attentional capacity and leads to a narrowing of the perceptual field causing a dehumanizing perspective of women as sexual objects for men's pleasure rather than individuals with thoughts and feelings, thereby increasing the propensity for sexual aggression. The present research also examines whether women's responses to this sexual objectification from men interfere with risk perception in sexual situations, particularly when women are drinking, increasing the likelihood of sexual victimization.

DETAILED DESCRIPTION:
These studies will provide a comprehensive test of our proposed model of alcohol-involved sexual assault that includes situation-specific mechanisms and key moderators of sexual violence. Specifically, hypotheses will be tested in the context of two carefully controlled laboratory studies. In Study 1, laboratory alcohol administration procedures will be used to manipulate intoxication (vs. placebo control) in men. Impaired attention and objectification will then be measured multi-modally including behavioral, self-report, and implicit measures. Finally, sexual aggression will be measured with a laboratory-based analogue of sexual assault. Study 2 will include women and follow the same alcohol administration procedures as Study 1. Additionally, mirroring men's objectification, objectifying gazes (vs. eye gazes) will also be manipulated. Impaired attention, self-objectification, and decreased sexual risk perceptions will then be assessed. Prior the laboratory visit, all participants will complete a battery of questionnaires to assess key moderators including a history of sexual assault perpetration and victimization, prior sexual objectification and self-objectification, as well as alcohol-related sex expectances and rape myth acceptance. The overall model will be analyzed within a conditional process model framework.

ELIGIBILITY:
Inclusion Criteria:

* 21-30 years of age
* at least social drinkers
* single
* men attracted to women, women attracted to men

Exclusion Criteria:

* current/past alcohol dependence (as assessed by a score of 8 or higher on the Alcohol Dependence Scale), alcohol-related treatment, or hospitalization due to alcohol use
* any past serious head injuries (as indicated by HELPS Brain Injury Screening Tool)
* serious psychological symptoms (defined as past psychotic, paranoid, or bipolar disorders, or current major depression)
* abstinence from alcohol use
* a condition or medication use in which alcohol consumption is medically contraindicated
* any legal restriction against drinking (e.g., as condition of probation or parole)
* presence of a positive breath alcohol concentration (BAC) upon arrival to the laboratory
* if the participant is less than six feet tall and weighs over 250 pounds or is over six feet tall and weighs over 300 pounds
* if a female participant is pregnant

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants who self-identify as men will participate in Study 1 and participants who self-identify as women will participant in Study 2
Enrollment: 359 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Laboratory analogue of sexual aggression | 20 minutes post alcohol or placebo dosing
  After learning that a woman does not like sexual media, male participants choose to show her a sexually explicit video or control video (selection of the sexually explicit video indicates more sexual aggression)
Sexual assault vignette measure of risk perception | 20 minutes post alcohol or placebo dosing
  Female participants read 18 vignettes describing a sexual interaction between a man and a woman that gets progressively riskier for sexual assault and indicate when they would leave the interaction (scores range from 1-18 and higher scores indicate worse risk perception)

SECONDARY OUTCOMES:
Eye-tracking measure of sexual objectification | 2 minutes post alcohol or placebo dosing
  Male participants wear a portable eye tracker and discuss media preferences with a female confederate while dwell time on the female confederate's face and body is monitored (longer dwell times on the woman's body and shorter dwell times on the woman's face indicate more sexual objectification)
Eye-tracking measure of self-objectification | 2 minutes post alcohol or placebo dosing
  Female participants wear a portable eye tracker and interact with a male confederate in front of a mirror while dwell time on the participant's body is monitored (longer dwell times on the participant's body indicates more self-objectification)
Object brief-implicit association task | 25 minutes post alcohol or placebo dosing
  On a computer, male participants sort stimuli words representing the categories object (e.g., tool), human (e.g., person), women (e.g., female), and men (male). Participants must respond as quickly and accurately as possible to categorize the words on a computer screen to object, human, women, and men categories via a computer key press. Responding faster to object and woman words and slower to woman and human words indicates implicit objectification of women
Self-object brief-implicit association task | 25 minutes post alcohol or placebo dosing
  On a computer, female participants sort stimuli words representing the categories object (e.g., tool), human (e.g., person), me (e.g., self), and others (them). Participants must respond as quickly and accurately as possible to categorize the words on a computer screen to object, human, me, and others categories via a computer key press. Responding faster to object and me words and slower to human and me words indicates implicit self-objectification.
Self-report state mindful attention awareness scale | 30 minutes post alcohol or placebo dosing
  Male and female participants self-report how attentive they feel on a 0 to 6 point scale (averaged lower scores indicate more mindful attention awareness)
Self-report other-objectification questionnaire | 35 minutes post alcohol or placebo dosing
  Male participants self-report how frequently they objectified the female confederate on a 1 to 6 point scale (averaged higher scores indicate more other-objectification)
Self-report self-objectification questionnaire | 35 minutes post alcohol or placebo dosing
  Female participants self-report how important appearance related attributes (e.g., sex appeal) are important to their self-concept relative to non-appearance attributes (e.g., hobbies) on a 0 to 9 point scale. Appearance attributes and non-appearance attributes are separately summed and non-appearance attribute scores are subtracted from appearance attribute scores (higher scores indicate more self-objectification)
Saliva collection | 5 minutes pre alcohol or placebo dosing, 5 minutes post alcohol dosing, and 20 minutes post alcohol or placebo dosing
  Female participants provide saliva samples to assess cortisol associated with stress responses

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Gervais, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data may be shared with other researchers (e.g., posted to the Open Science Framework) to aid with reproducibility and replicability of science.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified data may be made available to interested researchers when papers based on that data are published in scientific journals.
Access Criteria: Interested researchers will be required to have an Open Science Framework account.

DOCUMENTS (2):
  • Study Protocol (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03956238/Prot_005.pdf
  • Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT03956238/SAP_002.pdf